CLINICAL TRIAL: NCT03203070
Title: Laparoscopic-guided Transversus Abdominis Plane (TAP) Block for Postoperative Pain Control in Patients Undergoing Laparoscopic Roux-en-Y Gastric Bypass
Brief Title: Laparoscopic-guided TAP Block in Patients Undergoing Gastric Bypass
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Head of Department of Research in Bariatric Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HRJC/2017/17
Record Dates: First submitted 2017-06-25; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — metamizole magnesium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient and nursery staff evaluating postoperative pain do not know the applied intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metamizol iv (Active Comparator): The patients will receive only intravenous analgesia with Metamizole 2g/8 hours for control of postoperative pain.
  Interventions: Drug: Metamizol iv
- TAP block (Experimental): The patients will receive intravenous analgesia with Metamizol iv 2g/8h and intraoperative laparoscopic-guided TAP block for control of postoperative pain.
  Interventions: Drug: Metamizol iv; Procedure: TAP block

INTERVENTIONS:
Drug: Metamizol iv — Postoperative analgesia iv with Metamizol 2g/8h will be administered.
  Other Names: Nolotil
Procedure: TAP block — Intraoperative laparoscopic-guided TAP block will be performed with 30ml Bupivacaine 0.5%
  Other Names: Transversus abdominis plane block
  Arms: TAP block

SUMMARY:
A prospective randomized trial will be performed. Patients undergoing gastric bypass will be randomized into 2 groups: patients undergoing laparoscopic-guided transversus abdominis plane (TAP) block as part of multimodal analgesia (Group 1), associated with postoperative intravenous analgesia, and patients receiving only postoperative intravenous analgesia (Group 2).

Postoperative pain will be assessed with a Visual Analogic Scale 24h after surgery and morphine needs will be quantified.

DETAILED DESCRIPTION:
A prospective randomized trial will be performed. Patients undergoing laparoscopic Roux-en-Y gastric bypass will be randomized into 2 groups: patients undergoing laparoscopic-guided TAP block with 30 ml Bupivacaine 0.5%, as part of multimodal analgesia (Group 1), associated with postoperative intravenous analgesia (Metamizol 2g/8h and Acetaminophen 1g/8h), and patients receiving only postoperative intravenous analgesia (Metamizol 2g/8h and Acetaminophen 1g/8h) (Group 2).

Postoperative pain will be assessed with a Visual Analogic Scale 24 hours after surgery and morphine needs will be quantified.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >40 Kg/m2
* BMI >35 Kg/m2 and obesity associated comorbidities
* Patients undergoing laparoscopic Roux en Y gastric bypass

Exclusion Criteria:

* Patients undergoing other bariatric procedures, different than Roux en Y gastric bypass
* Patients undergoing open bariatric surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours after surgery
  Pain quantification will be assessed with a Visual Analogic Scale

CONTACTS AND LOCATIONS:
Overall Officials: Manule Duran, Study Director — Hospital Universitario Rey Juan Carlos
Locations (1):
- General Hospital Elche, Elche, Alicante, Spain

REFERENCES:
- [Derived] Ruiz-Tovar J, Garcia A, Ferrigni C, Gonzalez J, Levano-Linares C, Jimenez-Fuertes M, Llavero C, Duran M. Laparoscopic-Guided Transversus Abdominis Plane (TAP) Block as Part of Multimodal Analgesia in Laparoscopic Roux-en-Y Gastric Bypass Within an Enhanced Recovery After Surgery (ERAS) Program: a Prospective Randomized Clinical Trial. Obes Surg. 2018 Nov;28(11):3374-3379. doi: 10.1007/s11695-018-3376-8. PMID 29980989